CLINICAL TRIAL: NCT04445298
Title: Skin Barrier Assessment in Pregnancy and at Birth
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Jewish Health (Other)
Responsible Party: Sponsor
Other Study IDs: HS3513
Record Dates: First submitted 2020-04-29; First posted 2020-06-24 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Pregnancy Related; Allergy; Atopic Dermatitis Eczema; Asthma in Children; Food Allergy
MeSH Terms: conditions — Hypersensitivity; Food Hypersensitivity | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will obtain blood to assess the filaggrin gene mutation status, as filaggrin gene mutations have been associated with increased atopic dermatitis severity and persistence.
  Other blood work includes total immunoglobulin E and vitamin D.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pregnant women with expected delivery in the fall or winter: We will enroll up to 40 women who are expected to deliver in the fall (September, October, November) and winter (December, January, February). We will then follow their infant offspring.
  Interventions: Diagnostic Test: Transepidermal water loss; Diagnostic Test: Skin tape stripping; Diagnostic Test: Blood draw; Diagnostic Test: Bacterial PCR swab
- Pregnant women with expected delivery in the spring or summer: We will enroll up to 40 women who are expected to deliver in the spring (March, April, May) and summer (June, July, August). We will then follow their infant offspring.
  Interventions: Diagnostic Test: Transepidermal water loss; Diagnostic Test: Skin tape stripping; Diagnostic Test: Blood draw; Diagnostic Test: Bacterial PCR swab
- Infants born in the fall or winter: The infants born to the enrolled mothers will be followed. These are infants born in the fall (September, October, November) or winter (December, January, February).
  Interventions: Diagnostic Test: Transepidermal water loss; Diagnostic Test: Skin tape stripping; Diagnostic Test: Blood draw; Diagnostic Test: Bacterial PCR swab
- Infants born in the spring or summer: The infants born to the enrolled mothers will be followed. These are infants born in the spring (March, April, May) or summer (June, July, August).
  Interventions: Diagnostic Test: Transepidermal water loss; Diagnostic Test: Skin tape stripping; Diagnostic Test: Blood draw; Diagnostic Test: Bacterial PCR swab

INTERVENTIONS:
Diagnostic Test: Transepidermal water loss — We will assess the skin with transepidermal water loss (TEWL) by using a condenser-chamber system placed lightly on the skin. This will be performed at baseline, then after every 4 skin tape strips.
  Other Names: TEWL
Diagnostic Test: Skin tape stripping — Adhesive skin sampling discs will be pressed against the skin in a hairless location followed by lifting it free of the skin. The discs will be evaluated for lipid content, protein, and filaggrin byproducts in the collected skin sample.
  Other Names: STS
Diagnostic Test: Blood draw — We will draw blood to look at the vitamin D, total immunoglobulin E (IgE), and the filaggrin gene which is important in maintaining the skin barrier.
Diagnostic Test: Bacterial PCR swab — Skin swab from the superficial skin will be collected to be assessed in the laboratory via PCR for the presence of staphylococcus aureus.
  Other Names: PCR

SUMMARY:
This is a prospective birth cohort study assessing the role of maternal and environmental factors on the development of allergic diseases in children. Pregnant mothers will be enrolled and we will examine her skin barrier with skin tape strips (STS) and transepidermal water loss (TEWL), along with blood work. We will then follow her offspring and perform similar testing, along with detailed questionnaires inquiring about exposures such as use of detergents and soaps, sunlight exposure, and pollution exposure. When the infant is around 12 months old, we will contact the family via telephone to see if the child developed any allergic conditions within their first year of life, such as eczema, food allergy, or wheezing. A final questionnaire will be performed.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria of the pregnant women:

• Pregnant women at any stage of a singleton pregnancy.

Inclusion criteria of the infant:

• Infant is the offspring of a woman enrolled in the study.

Exclusion Criteria:

Exclusion criteria of all subjects:

* Use of systemic immunosuppressive drugs including oral steroids within 30 days of skin barrier assessment
* Has received total body phototherapy (e.g., ultraviolet light B [UVB], psoralen plus ultraviolet light A [PUVA], tanning beds [>1 visit per week]) within 30 days of skin barrier assessment
* Use of topical corticosteroids, topical immunomodulatory agents, or topical antibiotics on the extremity being evaluated within 7 days of skin barrier assessment
* Use of systemic antibiotics, antiparasitics, antivirals, or antifungals within 7 days, or antihistamines within 5 days of skin barrier assessment
* Has taken a bleach bath within 7 days of skin barrier assessment
* Use of emollients on the extremity being evaluated within 24 hours of skin barrier assessment
* Has taken a bath or shower on the day of the skin barrier assessment

Exclusion criteria of the pregnant women:

* Pregnant women with high risk pregnancies.
* Pregnancy is from an egg donation.
* Pregnant women pregnant with more than one fetus.
* Pregnant women with psychiatric and developmental co-morbidities that would render them unable to provide informed consent or perform study-related procedures.
* AIDS and HIV infection.
* A fetus with chromosomal or congenital abnormalities, a heritable hematological disorder like thalassemia or sickle cell disease in the mother.

Exclusion criteria of the infant:

* Infant is delivered earlier than 34 weeks gestation.
* Infant is born with a significant birth defect or medical condition where enrollment in this study is not in the infant's best interest.

Ages: 0 Minutes to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: We will enroll up to 40 pregnant mothers who are expected to deliver in the fall and winter, along with up to 40 pregnant mothers who are expected to deliver in the spring and summer. The infants will then be enrolled and followed in the study.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2020-08-03 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Skin barrier assessment with transepidermal water loss (TEWL) will be done in every infant. | 1 year
  TEWL will be performed in all infants to compare skin barrier assessments between infants born in the fall and winter with those born in the spring and summer. We hypothesize greater skin barrier dysfunction in those born in the fall and winter.
Skin barrier assessment with skin tape stripping (STS) will be done in every infant. | 1 year
  STS will be performed in all infants to compare skin barrier assessments between infants born in the fall and winter with those born in the spring and summer. We hypothesize greater skin barrier dysfunction in those born in the fall and winter.
Skin barrier assessment with skin swabs for staphylococcus aureus colonization will be done in every infant. | 1 year
  Skin swabs for staphylococcus aureus colonization will be performed in all infants to compare skin barrier assessments between infants born in the fall and winter with those born in the spring and summer. We hypothesize greater staphylococcus aureus colonization in those born in the fall and winter.
Skin barrier assessment with TEWL will be performed in every pregnant female and compared to her infant offspring, as well as between other pregnant females giving birth in other seasons. | 1 year
  We will compare the mother's skin barrier with the infant skin barrier to see if there is an association with the mother's skin barrier during pregnancy. We will perform TEWL to assess the degree of water loss before, during, and after skin tape stripping.
Skin barrier assessment with STS will be performed in every pregnant female and compared to her infant offspring, as well as between other pregnant females giving birth in other seasons. | 1 year
  We will compare the mother's skin barrier with the infant skin barrier to see if there is an association with the mother's skin barrier during pregnancy. We will perform STS to determine the skin breakdown products.
Skin barrier assessment with skin swabs for staphylococcus aureus colonization will be performed in every pregnant female and compared to her infant offspring, as well as between other pregnant females giving birth in other seasons. | 1 year
  We will compare the mother's skin barrier with the infant skin barrier to see if there is an association with the mother's skin barrier during pregnancy. We will perform skin swabs for staphylococcus aureus colonization to determine the presence of colonization.
Skin barrier assessment with filaggrin gene mutation status will be determined in everyone enrolled, and we will look for the filaggrin gene mutation in both the mother and infant. | 1 year
  The filaggrin gene is important for skin health, and we will assess for common filaggrin gene mutations in everyone enrolled in this study via a blood draw in the mother's and cord blood in the infants.
Vitamin D levels will be obtained and compared between individuals enrolled in this study. | 1 year
  Vitamin D levels will be obtained by blood draw in the pregnant mother's and cord blood in the infants. We will compare the values according to season of birth, as we hypothesize that the infants born in the fall and winter, along with their mothers, will have a lower vitamin D level.
Questionnaires regarding exposures will be compared with the skin barrier measurements to understand exposures that lead to increased skin barrier dysfunction. | 1 year
  Questionnaires will be administered to capture exposures during pregnancy, such as detergents, soaps, medications, and sunlight exposure. The answers will be compared with the results of the skin barrier assessment in both pregnant women and their infants to understand which exposures lead to skin barrier dysfunction.
Questionnaires and a follow up telephone call will allow us to see if infants born in the fall and winter have a higher incidence of allergy development. | 1 year
  Questionnaires and follow up telephone calls when the infant is 12 months old will determine which infants develop allergic conditions, such as atopic dermatitis, food allergy, and wheezing. We will compare the infants born in the fall and winter with those born in the spring and summer to see whether the infants born in the fall and winter have increased risk of developing allergy.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Leung, MD PhD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided